CLINICAL TRIAL: NCT04094571
Title: Characterizing the Delayed Muscle Response to Electrical Stimulation
Brief Title: Muscle Delay Characterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Science Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201901676 -N; 1762829 (Other Grant/Funding Number: National Science Foundation)
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Neurological Disorders
Keywords: functional electrical stimulation; rehabilitation
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Individuals and those with Movement Disorders (Experimental): Participants will perform the FES cycling protocol along with the FES angle protocol.
  Interventions: Device: Functional Electrical Stimulation (FES) Control Protocol; Device: Functional Electrical Stimulation (FES) Angle Protocol

INTERVENTIONS:
Device: Functional Electrical Stimulation (FES) Control Protocol — To measure the delay, the motor will take the tricycle crank to pre-specified angles and then hold that position while various combinations of the quadriceps femoris and the gluteal muscle groups are stimulated in study participants.
  Other Names: FES modified TerraTrike Rover recumbent tricycle
Device: Functional Electrical Stimulation (FES) Angle Protocol — To determine the effect of the crank angle on the FES delay and the muscle control effectiveness, the crank is positioned at a pre-specified angle, with various muscle groups being stimulated while holding this position. The motor then takes the crank to another angle and the process is repeated.
  Other Names: FES modified TerraTrike Rover recumbent tricycle

SUMMARY:
Functional electrical stimulation (FES) induced cycling is a common rehabilitative therapy. Closed-loop FES control holds the promise to improve rehabilitation procedures. However, FES results in a delay between the time of stimulation and muscle contraction and rapidly fatigues muscle. The purpose of this study is to measure the FES-induced delay on an FES cycle and to understand how the delay varies as a function of how long the user has been cycling and a function of the crank angle.

DETAILED DESCRIPTION:
This study will use non-invasive approaches (surface electrodes, encoders, torque meters, motors) to study muscle delay and how muscle fatigues for both individuals possessing movement disorders and healthy individuals. Individuals with movement disorders are often susceptible to partial or total paralysis. This paralysis often leads to an increasingly sedentary lifestyle. By implementing the intelligent closed-loop control of FES-cycling, FES-therapy can be made more effective, combating the effects of sedentary lifestyles. Using data obtained from non-invasive sensors, the study team will apply analytical techniques to quantify FES muscle delay and how well individuals can track a desired cadence as the muscle fatigues. A challenge associated with FES-induced cycling is that there exists a delay between the time when FES is applied and the time when the muscle contracts. There is likewise a delay between the time FES is removed and the time the muscle ceases to contract. Previous studies have measured this delay and determined that it varies with fatigue. A goal of this project is to measure this delay on an FES-cycle and to determine how this delay varies as a result of FES-induced cycling. Another goal is to determine what effect the crank angle has on the delay as well as on the muscle control effectiveness. This study will provide insight into how engineering can be combined with healthcare and therapy to better both fields and bridge the gap between engineering and medicine.

ELIGIBILITY:
Inclusion Criteria:

* healthy normal individuals aged 18-65 and individuals with movement disorders (e.g., spinal cord injury, Parkinson's disease, stroke)
* capable to perform the cycling exercises either voluntarily or under controlled electrical stimulation
* all participants have to be medically stable (i.e., do not exhibit asymptomatic osteoporosis, cardiopulmonary disease, pain, or other significant medical complications that would prohibit or interfere with testing or training)
* for neurologically impaired individuals, they should have a single neurologic condition
* under all situations the body size and weight of participant has to be compatible with the testing apparatus to ensure safety at all times

Exclusion Criteria:

* participants who are unresponsive to surface FES are not considered eligible for the study
* a history of significant cardiovascular disorders, chronic arterial diseases or congestive cardiac failure, including being medicated for hypertension and/or have an implanted pacemaker
* have a history of major musculoskeletal problems that limit hip and knee extension such as orthopedic surgery, including ACL reconstruction and/or joint replacements
* participants with denervated muscle, severe osteoporosis or abnormal bone formation in hip/knee joints, bone fractures, acute hernia, severe muscle spasticity, infection in the lower extremities, epilepsy, diabetes, severe angina, pressure ulcers, vein thrombosis, and any ailments causing high fever, high blood pressure or high heart rate
* pregnant women, children/minors, adults with diminished decision-making capacity, and non-English speakers
* under all situations the body size and weight of participant has to be compatible with the testing apparatus to ensure safety at all times

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Measure of crank torque | Day 1
  A torque meter (SRM Science PowerMeter) is attached to the tricycle's crank to provide instantaneous feedback of the rider torque. A combination of muscle groups will be stimulated and the resulting crank torque will be measured by the meter.

CONTACTS AND LOCATIONS:
Overall Officials: Warren Dixon, PhD, Principal Investigator — University of Florida
Locations (1):
- NCR lab in MAE-B building at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No